CLINICAL TRIAL: NCT05884632
Title: Daily Adaptive RadioTherapy in Postoperative HypofrActionated Salvage radiothERapy for Prostate Cancer Patients
Acronym: DART-PHASER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-51
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients will be treated on the prostate bed with Ethos using daily-adaptive modality with the dose of 59 Gy in 20 daily fractions of 2.95 Gy
  Interventions: Radiation: Daily Adaptive RadioTherapy

INTERVENTIONS:
Radiation: Daily Adaptive RadioTherapy — Patients will be treated on the prostate bed with Ethos using daily-adaptive modality with the dose of 59 Gy in 20 daily fractions of 2.95 Gy

SUMMARY:
This is a monoinstitutional prospective pilot study, aiming to evaluate treatment-related toxicity of an hypofractionated postoperative salvage radiotherapy with daily-adaptive modality in patients affected by prostate cancer biochemical recurrence.

Patients will be treated with postoperative hypofractionated salvage radiotherapy with a dose of 59 Gy in 20 fractions with daily-adaptive modality. Considering the consolidate role and clinical outcome of postoperative hypofractionated radiotherapy with elevate level of evidence (8-10), the study will not be controlled, but compared with literature data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 80 years;
* Prostate cancer diagnosis, pT2-3 pN0, any resection margin (R0 or R1);
* Indication to local salvage treatment defined as: early salvage radiotherapy after primary prostate surgery (radical prostatectomy) with PSA <0.2 ng/ml or salvage radiotherapy after primary prostate surgery (radical prostatectomy) with PSA ≥0.2 ng/ml;
* No distant metastases (M0) diagnosed with PSMA-PET-CT;
* Informed consent to trial's participation and personal data treatment.

Exclusion Criteria:

* Age <18 years old;
* Adjuvant radiotherapy;
* Previous radiation in the same anatomical site.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Acute gastrointestinal toxicity | 90 days from the RT treatment
  Will be evaluated by physician-reported outcome according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0) and by patient-reported outcome according to the EPIC questionnaire. More specifically, acute toxicity will be defined as any gastrointestinal event occurred within 90 days from the RT treatment with grade ≥G2.

SECONDARY OUTCOMES:
Acute genitourinary toxicity | 90 days from the RT treatment.
  Will be evaluated by physician-reported outcome according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0), and by patient-reported outcome according to the EPIC questionnaire. More specifically, acute toxicity will be defined as any genitourinary event occurred within 90 days from the RT treatment.
Late toxicity | From 90 days after the RT treatment until 24 months
  Will be evaluated by physician-reported outcome according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0), and by patient-reported outcome according to the EPIC questionnaire. More specifically, late toxicity will be defined as any event (genitourinary and gastrointestinal) occurred from 90 days after the RT treatment.
QLQ-C30 | At screening, 2nd and 4th week during RT, at 3, 6, 12, and 24 months
  Patient-reported outcomes will be assessed via the EORTC global (QLQ-C30) questionnaires at screening, 2nd and 4th week during RT, at 3, 6, 12, and 24 months
Biochemical failure | 24 months
  PSA raise after RT from nadir
Time to biochemical failure | 24 months
  Time between salvage RT and biochemical failure
Local in-field relapse | 24 months
  Local in-field relapse evaluated with PET-CT or RM
Metastases-free survival | 24 months
  Metastases-free survival evaluated with PSMA PET-TC in case of PSA raise

CONTACTS AND LOCATIONS:
Overall Officials: Luca Nicosia, Principal Investigator — IRCCS Sacro Cuore Don Calabria - Dipartimento di Radioterapia Oncologica Avanzata
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy